CLINICAL TRIAL: NCT03243227
Title: Effectiveness of Neurodynamic Techniques for the Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Hayat Hamzeh, Lecturer, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 47/2016/2256
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; neurodynamics; median nerve gliding exercise
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodynamic techniques (Experimental): 4 sessions of Neurodynamics treatment will be provided by an experienced physiotherapist. It will include manual therapy, median nerve gliding exercise, median nerve tension exercise. patients will continue the exercises as home exercise program during and after the treatment period.
  Interventions: Other: Neurodynamic techniques
- Exercise (Active Comparator): Exercise therapy 4 sessions of exercise treatment will be provided by an experienced physiotherapist. It will include active range of motion, stretching, and strengthening exercise. patients will be given a brochure to continue the exercises as home exercise program during and after the treatment period.
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Neurodynamic techniques — 4 sessions of Neurodynamics treatment will be provided by and experienced physiotherapist. It will include manual therapy, median nerve gliding exercise, median nerve tension exercise. patients will continue the exercises as home exercise program during and after the treatment period.
  Arms: Neurodynamic techniques
Other: Exercise therapy — AROM exercise stretching exercise strengthening exercise 4 sessions
  Arms: Exercise

SUMMARY:
Carpal tunnel syndrome CTS is the most common peripheral neuropathy seen in clinic. It results in marked functional limitations of patients. Most patients undergo surgical release which places a heavy burden on health system. Neurodynamic exercise is claimed to be an effective physiotherapy treatment for these patients. It is a practical and complications-free treatment which can be used as a home exercise program. This study aims to investigate the effect of median nerve gliding exercise on symptoms severity and functional limitation in CTS patients.

DETAILED DESCRIPTION:
* Design: Two groups randomized controlled trial
* Participants: 50 subjects diagnosed with CTS will be recruited from JUH physical medicine and rehabilitation department, diagnosis will be confirmed by a physician clinically and using nerve conduction test. Subjects will be randomized into treatment and control groups.
* Procedures: Participants will be recruited from the physical medicine department at JUH and the diagnosis and initial assessment will be performed by a physician. Baseline outcomes will be measured by an experienced physiotherapist.

Treatment Group: Neurodynamics evaluation and treatment will be provided by an experienced physiotherapist. Each treatment session involves both manual therapy and median nerve mobilization exercise following the neurodynamics concept. Four 60 minutes sessions over a period of four weeks will be performed for each patient. Median nerve mobilization exercise will be continued as home exercise program and will be monitored by the treating physiotherapist using exercise diary.

Control group: four sessions of exercise will be given to participants. CTS standard exercise brochure will be given for the patients to follow over 4 weeks. The brochure will include wrist joint strengthening, stretching and AROM exercise.

Outcomes will be measured at the end of the 4 weeks treatment, 6 weeks and 6 months post treatment.

• Data analysis: Microsoft Excel and SPSS will be used for data entry and analysis.

Descriptive analysis: All obtained data will be tabulated, means, standard deviations and differences will be measured.

Inferential analysis: Two way repeated measure ANOVA will be used to measure differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

Confirmed CTS diagnosis

Exclusion Criteria:

Previous trauma or surgery involving the upper extremities known neurological condition pregnancy history of radiating neck or back pain in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Boston Carpal Tunnel Questionnaire score | Baseline, 1 month, 6 months
  BCTS is a patient-based outcome measure used for patients with CTS. It includes two distinct scales, the Symptom Severity Scale (SSS) which has 11 questions and uses a five-point rating scale and the Functional Status Scale (FSS) containing 8 items which have to be rated for degree of difficulty on a five-point scale. Each scale generates a final score (sum of individual scores divided by number of items) which ranges from 1 to 5, with a higher score indicating greater disability.

SECONDARY OUTCOMES:
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | Baseline, 1 month, 6 months
  DASH is a patient-based outcome measure used to assess function in patients with arm or hand pain. it includes two components: the disability/symptom
Pain severity scale | Baseline,1 month , 6 months
  subjective rating of pain severity is specified by patient as a number from 0-10. the higher the number the greater level of pain
Wrist ROM | Baseline, 1 month , 6 months
  Range of movement of the wrist joint is measured using universal goniometer. All wrist joint movements will be measured actively and passively.
Grip strength | Baseline, 1 month, 6 months
  Hand grip strength is measured using a hand held dynamometer device. Reading is taken in pounds.
Surgery | 6 months
  whether or not the patient decided to undergo median nerve decompression surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hayat Hamzeh, MSC, Principal Investigator — Lecturer
Locations (1):
- The University of Jordan, Amman, Jordan